CLINICAL TRIAL: NCT07013344
Title: Association of Plasma N-terminal Pro-Brain Natriuretic Peptide Levels With the Burden of Coronary Artery Disease: Insights From a Real-World Cohort
Brief Title: Association of Plasma N-terminal Pro-Brain Natriuretic Peptide Levels With the Burden of Coronary Artery Disease
Acronym: BNP-CAD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Carlo Gaspardone, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: BNP-CAD-HSR-2025
Record Dates: First submitted 2025-03-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Coronary Syndrome; Chronic Coronary Total Occlusion; Coronary Arterial Disease (CAD); Stable Chronic Angina; NT-pro-BNP
Keywords: NT-pro-BNP; Coronary Arterial Disease (CAD); Chronic Coronary Syndrome (CCS)
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: BNP — Measurement of plasma NT-proBNP level.

SUMMARY:
This study aim to investigate the association between plasma NT-proBNP levels and the presence, extent and severity of stenosis in patients with suspected coronary artery disease.

DETAILED DESCRIPTION:
The investigators prospectively measured plasma NT-proBNP levels in consecutive patients referred to the center for elective diagnostic coronary angiography due to symptoms or signs of coronary artery disease over a two- year period. Patients with conditions known to elevate NT-proBNP levels, including heart failure, severe valvular disease, atrial fibrillation, severe chronic kidney disease (eGFR < 30 mL/min), prior coronary artery bypass grafting, or age over 80 years, were excluded.

ELIGIBILITY:
Inclusion Criteria:

* patient referred for elective coronary angiography due to suspected CAD.
* NT-proBNP measurement during hospitalization

Exclusion Criteria:

* heart failure
* severe valvular disease
* atrial fibrillation
* severe chronic kidney disease (eGFR < 30 mL/min)
* prior coronary artery bypass grafting
* age over 80 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to San Raffaele Hospital between September 2021 and July 2024 for elective coronary angiography due to the suspected CAD (i.e. presence of suggestive signs or symptoms and positive non-invasive functional and/or anatomical tests).
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Association between plasma NT-proBNP levels and the presence, extension and severity of angiographic lesions in patients with suspected CAD. | Plasma NT-proBNP levels are quantified on the morning before coronary angiography. The CAD burden is independently evaluated by two experienced interventional cardiologists periprocedurally and immediately after the coronary angiography.
  Plasma NT-proBNP levels are quantified on the morning before coronary angiography using a highly sensitive electrochemiluminescence immunoassay (ECLIA) method (NT-proBNP, Roche Diagnostics, Germany), employing the Roche Modular Analytics E170 immunoassay analyzer AL.
  The aim of this study is to explore the association between these levels and the presence (critical vs non-critical), location (prognostic vs non-prognostic), severity (>70%, 70-99%, 100%) and extent of obstructive lesions detected in a contemporary cohort of patients undergoing coronary angiography for suspected CAD. Coronary angiograms are independently evaluated by two experienced interventional cardiologists (C.G. and C.G.) who are blinded to the NT-proBNP levels.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy, Italy